CLINICAL TRIAL: NCT04809688
Title: Effects of Saskatoon Berry on Glucose Metabolism, Insulin Resistance and Gut Microbiota in Healthy Human Subjects
Brief Title: Saskatoon Berry on Metabolism and Gut Microbiota in Healthy Subjects
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Garry Shen, Dr. Gary Shen, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS23500 (B2019:122)
Record Dates: First submitted 2020-10-15; First posted 2021-03-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: Saskatoon berry; Glucose tolerance; Gut microbiota; Healthy subjects
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Healthy subject (n=20) will be enrolled in a single group for oral administration of dried Saskatoon berry as snack.
  Healthy subjects (n=10) will be enrolled in a single group for assessing glycemic index for dried Saskatoon berry.
  Prediabetes (n=20) will be randomized in two groups for dried Saskatoon berry and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm for healthy subjects using dried whole Saskatoon berry
  Interventions: Dietary Supplement: Saskatoon berry; Dietary Supplement: Dried Saskatoon berry

INTERVENTIONS:
Dietary Supplement: Saskatoon berry — Freeze dried Saskatoon berry (30 g) will be orally administrated daily for 10 weeks.
Dietary Supplement: Dried Saskatoon berry — Prediabetic patients (fasting glucose 5.6-6.9 mM/L, HbA1c 5.7-6.9%, or OGTT 2 h glucose 7.8-11 mM/L) will be randomized in two groups. One group participants will take 40g of dried Saskatoon berry/day for 12 weeks. Another group will take 40g of dried Saskatoon berry/day for 12 weeks,

SUMMARY:
Diabetes becomes epidemic in worldwide countries. Nine out of ten diabetic patients are type 2 diabetes (T2D). T2D is characterized by insulin resistance and obesity. Uncontrolled diabetes leads to serious consequences including heart attack, stroke, chronic renal failure, liver failure, blindness and low limb amputation. Most of hypoglycemic medications have side effects. Natural foods or nutraceuticals with hypoglycemic potential are expected to provide a safer management for diabetic patients. Saskatoon berry is a popular fruit in Canadian Prairie and Northern states in USA. Our recent studies demonstrated Saskatoon berry (SB) powder attenuated hyperglycemia, hyperlipidemia, insulin resistance, inflammation, liver steatosis and gut dysbiosis in diet-induced insulin resistant mice, a model for T2D. The results in anti-diabetic activities of SB powder have been supported by other groups in high fat fed rats. Our preliminary studies in 20 healthy subjects demonstrated that dried whole SB (40 g/day for 10 weeks) significantly reduced fasting plasma glucose, total and LDL-cholesterol, systolic blood pressure, and increased plasma glucagon-like peptide compared to baseline, which was associated with increased intake of total fiber and decreased intake of saturated fat. The changes in metabolic and vascular variables significantly correlated with the alterations in gut microbiota. The combination of findings suggest that Saskatoon berry is good candidate of prebiotic functional food as a supplemental remedy for reducing the risk for metabolic syndrome and preventing or managing T2D. The effect of Saskatoon berry and its products on metabolic disorders have not been studied in healthy human subjects. We propose to examine the effects of oral administration of freeze-dried whole SB on glucose metabolism, insulin resistance and gut microbiota in healthy subjects in a single arm, open labeled phase I clinical trial.

DETAILED DESCRIPTION:
Subject recruitment: Healthy subjects and prediabetes (males and females, 18-75 years of age) in Winnipeg, who are voluntarily signing an informed consent approved by Research Ethics Board in University of Manitoba, will be eligible to the study. Exclusion criteria include: 1) candidates have a history of myocardial infarction, stroke, hypertension, diabetes, hyperlipidemia, chronic kidney disease; 2) participants are taking hypoglycemic, anti-hypertensives, lipid lowering medications or antibiotics within a month.

Dietary product: Freeze dried Saskatoon berry have been obtained from Prairie Berries Inc. The berries were freshly frozen and no any supplementation was added to the dried berry. The product has been processed by certified facilities and the batch of dried berry has passed pathogen analysis.

Regimen: Participants (n=20) will orally administrate 30 g/day of freeze dried Saskatoon berry during breakfast for 10 weeks.

Scheduled visits:

Visit 1: Consent and enrollment. A questionnaire for domestic questionnaire including dietary intake and physical activity will be filled. Measurements of body weight, height and blood pressure will be taken during the visit.

Visit 2 (<1 week from the visit 1 and before the start of berry administration): 75 g oral glucose tolerance test (OGTT) after an overnight fasting. Insulin, glucagon-like peptide-1 (GLP-1), liver enzymes (alanine transaminase or ALT, aspartate transaminase or AST), creatinine, lipid profile and inflammation markers (high-sensitive C-reactive protein or hs-CRP) will be measured as baseline. Stool samples will be collected in stool DNA preservation and collection kit.

Participants will be provided with sealed packages of dried Saskatoon berry and instruction of the administration. Insulin and lipid profile will be tested in blood samples withdrawn at fast glucose for OGTT.

Visit 3 (at 5 weeks after the start of administration of Saskatoon berry): Participants will be asked to provide feedback on general well-being and the intake of Saskatoon berry. Body weight, blood pressure and heart rate will be measured and recorded.

Visit 4 (at 10 weeks after the start of the dietary regimen): Participants will be asked to collect stool sample with the collection kit within 1 week before the visit and bring it to the visit. They will also be asked to have an overnight fasting the night before visit. They will receive blood withdrawal for biochemical tests and OGTT as the same as visit 2. During the visit, body weight, blood pressure and heart rate of participants will be taken. Questionnaires on participants' dietary intake, physical activity and feedback to the study will be completed.

Participants will receive a $50 honorarium gift card for their participation. Sample collection and analyses: OGTT, ALT, AST, creatinine and lipid profile will be analyzed in Clinical Chemistry in Health Science Centre, Winnipeg. Insulin, hs-CRP and GLP-1 will be analyzed in the Dr. G. Shen's laboratory. Homeostatic model assessment-insulin resistance or homeostatic model assessment for insulin resistance (HOMA-IR) will be calculated based on fasting plasma glucose and insulin. Stool samples will be aliquoted and stored under -80°C before submission. Microbiome analysis will be conducted in Integrate Microbiome Resource at Dalhousie University. Fecal short chain fatty acids (SCFA) will be measured in Microbiome Insight in University of British Columbia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects living in Winnipeg.
2. Willingness to sign an informed consent.

Exclusion Criteria:

1. History of myocardial infarction, stroke, hypertension, diabetes, hyperlipidemia, chronic kidney disease.

2) Participants are taking hypoglycemic, anti-hypertensives, lipid lowering medications or antibiotics within a 1 month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | Changes from baseline to 10 weeks after the start of dietary intervention
  Fasting plasma glucose in mM/L
Total serum cholesterol | Changes from baseline to 10 weeks after the start of dietary intervention
  Fasting total cholesterol in mM/L

SECONDARY OUTCOMES:
Lipid profile beside total cholesterol | Onset and 10 weeks after the start of dietary intervention
  Triglycerides, LDL-cholesterol, HDL-cholesterol and non-HDL-cholesterol in mM/L
C-reactive protein | Onset and 10 weeks after the start of dietary intervention
  C-reactive protein in mg/L
Liver enzymes | Onset and 10 weeks after the start of dietary intervention
  ALT, AST in units/L
Body mass index accord to body weight and height | Onset, 5 and 10 weeks after the start of dietary intervention
  Body weight in kg, heights in cm, and body mass index in kg/M^2
Blood pressure | Onset, 5 and 10 weeks after the start of dietary intervention
  Systolic and diastolic blood pressure in mmHg
Gut micrbiota | Baseline and 10 weeks of SB intake
  16S-rRNA sequencing of stool samples
Glucagaon-like peptide | Between baseline and 10 weeks of SB intake
  Plasma levels analyzed using ELISA
Insulin and homeostasis model assessment of insulin resistance (HOMA-IR) | Between baseline and 10 weeks of SB intake
  Fasting plasma insulin analyzed using ELISA and HOMA-IR estimated via simultaneous plasma glucose and insulin

OTHER OUTCOMES:
Dietary intake, physical activities | Onset and 10 weeks after the start of dietary intervention
  3 day food intake and the type in gram, frequency in time/day and length of physical activities index in artificial score (score scale 0-3, high means more activity)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Shen, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao R, Khafipour E, Sepehri S, Huang F, Beta T, Shen GX. Impact of Saskatoon berry powder on insulin resistance and relationship with intestinal microbiota in high fat-high sucrose diet-induced obese mice. J Nutr Biochem. 2019 Jul;69:130-138. doi: 10.1016/j.jnutbio.2019.03.023. Epub 2019 Apr 9. PMID 31078906
- [Background] Huang F, Zhao R, Xia M, Shen GX. Impact of Cyanidin-3-Glucoside on Gut Microbiota and Relationship with Metabolism and Inflammation in High Fat-High Sucrose Diet-Induced Insulin Resistant Mice. Microorganisms. 2020 Aug 14;8(8):1238. doi: 10.3390/microorganisms8081238. PMID 32824001
- [Background] du Preez R, Wanyonyi S, Mouatt P, Panchal SK, Brown L. Saskatoon Berry Amelanchier alnifolia Regulates Glucose Metabolism and Improves Cardiovascular and Liver Signs of Diet-Induced Metabolic Syndrome in Rats. Nutrients. 2020 Mar 27;12(4):931. doi: 10.3390/nu12040931. PMID 32230955